CLINICAL TRIAL: NCT02664116
Title: IM Ketorolac vs Diclofenac Potassium Powder for Oral Solution (Cambia) for the Acute Treatment of Severe Migraine
Brief Title: IM Ketorolac vs Cambia for the Acute Treatment of Severe Migraine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Health (Other)
Collaborators: Depomed (Industry)
Responsible Party: Principal Investigator, Emily Rubenstein Engel, Associate Director, Dalessio Headache Center, Scripps Clinic, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHC-002
Record Dates: First submitted 2016-01-18; First posted 2016-01-26 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Headache
Keywords: Severe Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Solutions; Diclofenac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cambia (Experimental): Diclofenac postassium powder for oral solution and placebo injection
  Interventions: Drug: Diclofenac postassium powder for oral solution and placebo injection
- ketorolac (Active Comparator): ketorolac intramuscular injection and placebo oral solution
  Interventions: Drug: Ketorolac intramuscular injection and placebo oral solution

INTERVENTIONS:
Drug: Diclofenac postassium powder for oral solution and placebo injection — Diclofenac postassium powder for oral solution 50 mg in 1 ounce water orally, single dose and placebo normal saline 2ml intramuscular injection, single dose
  Other Names: Cambia
  Arms: Cambia
Drug: Ketorolac intramuscular injection and placebo oral solution — ketorolac 60 mg in 2 ml intramuscular injection, single dose and placebo oral solution, 1 ounce, single dose
  Other Names: Toradol
  Arms: ketorolac

SUMMARY:
This research will be conducted to see if the oral drug Cambia is as effective in relieving severe migraine headaches as the injectable drug ketorolac.

DETAILED DESCRIPTION:
The treatment of severe migraine often requires a patient office visit or treatment in the ER or urgent care setting. This is due to the minimal efficacy of PO treatments once migraine is severe, and therefore the need for parenteral treatments. IM Ketorolac is one mainstay of parenteral treatment. There is an unmet need for effective at-home treatment regimens for severe migraine. Despite FDA approval of Cambia for acute migraine treatment, insurance is reticent to cover the treatment due to higher cost in comparison to generic diclofenac tablets, despite superior efficacy of Cambia in comparison to generic diclofenac tablets (Diener, Cephalalgia 2006). One objective of this study would be to provide rationale to justify the insurance coverage of this treatment in comparison to generic tablets, because at home treatment is less costly than office visit or emergency department visit to receive IM ketorolac.

A previous study of Cambia demonstrated that this formulation of diclofenac potassium for oral solution is effective in reducing pain intensity within 30 minutes, which may be related to the 15-minute Tmax associated with this formulation. The rapid-onset benefits were sustained through 24 hours post-treatment (Lipton, Cephalalgia 2010)

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet IHS criteria for migraine
* Age 18 to 65
* At least 2 migraine attacks per month
* Able to give written consent
* Willing to complete the entire course of the study
* Current headache duration greater than or equal to 36 hours

Exclusion Criteria:

* Pregnant or nursing
* Significant medical or psychiatric disease
* History of gastritis, gastric ulcer, GI bleed
* Renal insufficiency
* Hepatic insufficiency
* History of opioid dependence within the last 10 years or currently
* Any current or prior use of DICLOFENAC POTASSIUM POWDER FOR ORAL SOLUTION (CAMBIA)
* Past allergic reaction to DICLOFENAC or other NSAIDs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pain relief, 0-3 scale | Change from baseline pain rating at 5, 10, 15, 30, and 60 minutes post intervention
Pain free response, 0-3 scale | 2 hours post intervention
Sustained pain free response, 0-3 scale | 24 hours post intervention

SECONDARY OUTCOMES:
Change in severity of migraine associated symptoms | 5, 10, 15, 30, 60, 120 minutes and 24 hours post intervention
  Disability, Nausea, Photophonia/phonophobia self reported using a 0-3 rating scale
Return to function | 24 hours post intervention
  Severity, Disability, Nausea, Photophonia/phonophobia self reported as 0 on 0-3 scale

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rubenstein Engel, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data will not be made available

REFERENCES:
- [Background] Factor SA, Jankovic J. Randomized trial of IV valproate vs metoclopramide vs ketorolac for acute migraine. Neurology. 2014 Oct 7;83(15):1388-9. doi: 10.1212/01.wnl.0000455698.16732.0a. No abstract available. PMID 25288700
- [Background] Garnock-Jones KP. Diclofenac potassium powder for oral solution: a review of its use in patients with acute migraine. CNS Drugs. 2014 Aug;28(8):761-8. doi: 10.1007/s40263-014-0186-y. PMID 25034250
- [Background] Friedman BW, Garber L, Yoon A, Solorzano C, Wollowitz A, Esses D, Bijur PE, Gallagher EJ. Randomized trial of IV valproate vs metoclopramide vs ketorolac for acute migraine. Neurology. 2014 Mar 18;82(11):976-83. doi: 10.1212/WNL.0000000000000223. Epub 2014 Feb 12. PMID 24523483
- [Background] Taggart E, Doran S, Kokotillo A, Campbell S, Villa-Roel C, Rowe BH. Ketorolac in the treatment of acute migraine: a systematic review. Headache. 2013 Feb;53(2):277-87. doi: 10.1111/head.12009. Epub 2013 Jan 8. PMID 23298250
- [Background] Lipton RB, Grosberg B, Singer RP, Pearlman SH, Sorrentino JV, Quiring JN, Saper JR. Efficacy and tolerability of a new powdered formulation of diclofenac potassium for oral solution for the acute treatment of migraine: results from the International Migraine Pain Assessment Clinical Trial (IMPACT). Cephalalgia. 2010 Nov;30(11):1336-45. doi: 10.1177/0333102410367523. Epub 2010 Apr 7. PMID 20959428
- [Background] Duarte C, Dunaway F, Turner L, Aldag J, Frederick R. Ketorolac versus meperidine and hydroxyzine in the treatment of acute migraine headache: a randomized, prospective, double-blind trial. Ann Emerg Med. 1992 Sep;21(9):1116-21. doi: 10.1016/s0196-0644(05)80654-7. PMID 1514724
- [Background] Orr SL, Aube M, Becker WJ, Davenport WJ, Dilli E, Dodick D, Giammarco R, Gladstone J, Leroux E, Pim H, Dickinson G, Christie SN. Canadian Headache Society systematic review and recommendations on the treatment of migraine pain in emergency settings. Cephalalgia. 2015 Mar;35(3):271-84. doi: 10.1177/0333102414535997. Epub 2014 May 29. PMID 24875925
- [Background] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Background] Diener HC, Montagna P, Gacs G, Lyczak P, Schumann G, Zoller B, Mulder LJ, Siegel J, Edson K. Efficacy and tolerability of diclofenac potassium sachets in migraine: a randomized, double-blind, cross-over study in comparison with diclofenac potassium tablets and placebo. Cephalalgia. 2006 May;26(5):537-47. doi: 10.1111/j.1468-2982.2005.01064.x. PMID 16674762
- [Derived] Engel ER, Cheng J. IM ketorolac vs diclofenac potassium powder for oral solution for the acute treatment of severe migraine: a randomized controlled trial. Neurol Sci. 2020 Mar;41(3):537-542. doi: 10.1007/s10072-019-04157-y. Epub 2019 Dec 12. PMID 31833000